CLINICAL TRIAL: NCT03783663
Title: Sleep Self-management in Pregnancy Using a Personalized Health Monitoring Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Amherst (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2017-3846
Record Dates: First submitted 2018-12-17; First posted 2018-12-21 (Actual); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Pregnancy; Sleep

STUDY DESIGN:
Intervention Model Description: parallel arm superiority, pilot feasibility randomized controlled trial
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep education plus Misfit Shine 2 (Experimental): This arm receives sleep education from the study nurse and also receives a Misfit Shine 2 to wear for 12 weeks to self-monitor sleep.
  Interventions: Behavioral: Misfit Shine 2
- sleep education only (No Intervention): This arm receives only sleep education from the study nurse.

INTERVENTIONS:
Behavioral: Misfit Shine 2 — The intervention group was given a Misfit Shine 2 to monitor sleep throughout the 12-week intervention period. Participants were instructed to wear the device on the wrist, which is better for capturing sleep than the other wear locations. Participants were instructed on how to self-monitor total sleep time and select a goal for that behavior. Further, participants were asked to view feedback on their sleep time daily on the Misfit smartphone app, which they used to monitor their progress toward achieving their behavioral goals.
  Arms: Sleep education plus Misfit Shine 2

SUMMARY:
Pregnancy-associated sleep disorders are a common acute experience in pregnancy experienced by up to 82% of women. Sleep disorders are associated with increased risk for pre-eclampsia, gestational diabetes, longer labor, cesarean birth, and postpartum depression, and are higher among pregnant women of lower socioeconomic status. Traditional clinical management of sleep disorders in pregnancy includes education and counseling on sleep hygiene and sleep positioning, dietary modifications, relaxation, iron supplementation, weight management, and physical activity, yet education-based behavioral interventions show minimal effectiveness for improving sleep among pregnant women. These methods typically do not incorporate objective self-monitoring, which is an important behavior change technique. In pregnancy, objective self-monitoring on a day-to-day basis is particularly important as sleep disorders may worsen as pregnancy progresses.

Computer-based personalized health monitoring (PHM) devices may serve as an effective tool with which pregnant women can self-manage sleep through incorporation of regular feedback. This strategy may be beneficial not only for women with pregnancy-associated sleep disorders but also for pregnant women with less severe sleep disruptions that experience daytime sleepiness, fatigue, and decreased quality of life. PHM devices have been used to promote weight loss, diet, and physical activity changes but no studies have specifically targeted sleep among pregnant women. The purpose of this pilot study is to establish the feasibility and acceptability of conducting a 12-week intervention for sleep self-management with pregnant women using a PHM device, in order to refine the intervention for a larger, randomized trial.

ELIGIBILITY:
Inclusion Criteria: at time of recruitment (t0) women must:

1. be age ≥ 18
2. 14 to <24 completed weeks gestation of pregnancy

2) have no known maternal or fetal complications 3) have a smartphone compatible with the study PHM device 4) have internet access 5) be English speaking 6) be receiving prenatal care.

Exclusion Criteria:

1. pre-existing diabetes mellitus or hypertension
2. diagnosed sleep disorder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-07-18 (Actual); Study Completion 2018-08-27 (Actual)

PRIMARY OUTCOMES:
Number of participants that remain in the study for the entire study period for the intervention and control groups. | 24 to 36 weeks gestation of pregnancy
  To assess feasibility of the study, we will calculate the number and percentage of participants in both groups that remain in the study for the entire study period. The study will be considered as feasible if at least 80% of participants remain in the study for its entirety.
Percentage of days during which the Misfit Shine 2 is worn by participants in the intervention group. | 24 to 36 weeks gestation of pregnancy
  To assess feasibility of the study, for women in the intervention group, we will calculate the proportion of the number of days the Misfit Shine 2 is worn during the study period. We will consider the intervention as feasible if participants wear the Misfit Shine 2 at least 80% of days during the study period.
Participant satisfaction with the sleep education (both groups) and with the Misfit Shine 2 (intervention group only) will be assessed through qualitative interviews. | 36 weeks gestation of pregnancy.
  At 36 weeks gestation, all participants will be asked to take part in a semi-structured qualitative interview in which open-ended questions will be asked about their sleep patterns, barriers and facilitators of sleep, and whether the sleep education was deemed helpful. Intervention group participants will additionally be asked questions about the experience wearing the MisFit Shine 2, their like and dislikes, and whether they believe it would be helpful to other pregnant women.

SECONDARY OUTCOMES:
Sleep quality and duration as measured by the Pittsburgh Sleep Quality Index (PSQI) | 24 to 36 weeks gestation of pregnancy
  The PSQI is a 19-item survey questionnaire measuring perceived sleep quality and disturbance over the past month. It has been used in numerous studies with pregnant women and has been validated for pregnant women using confirmatory factor analysis and has reliability of .7460. Scores ≥ 5 will be considered indicative of poor sleep.
Sleep disturbances as measured by the PROMIS SF v1.0-Sleep Distrubance 6a | 24 to 36 weeks gestation of pregnancy
  The PROMIS SF v1.0-Sleep Distrubance 6a is a validated 6-item survey questionnaire that measures individual perceptions of sleep quality and disturbance in the past seven days using a 5-point Likert scale. It is scored by summing responses for all items (two are reverse scored); higher scores indicate higher sleep disturbance.
Excessive daytime sleepiness as measured by the Epworth Sleepiness Scale | 24 to 36 weeks gestation of pregnancy
  The Epworth Sleepiness Scale is an 8-item survey questionnaire of daytime sleepiness. It has been validated for measuring symptoms of daytime sleepiness in pregnant women using principal components and confirmatory factor analysis, and has a reliability coefficient of 0.75. Higher cumulative scores indicate higher sleepiness.
Fatigue as measured by the PROMIS Fatigue Short Form 4a | 24 to 36 weeks gestation of pregnancy
  This 4-item survey questionnaire measures fatigue in the past seven days with a 5-point Likert scale. Responses for all items are summed; higher scores indicate higher fatigue symptoms.
Depressive symptoms as measured by the PROMIS Depression Short Form 6a and the Edinburgh Postnatal Depression Scale | 24 to 36 weeks gestation of pregnancy
  The PROMIS Depression Short Form 6a is a 6-item survey questionnaire that measures depressive symptoms in the past seven days using a 5-point Likert scale. It is scored by summing the responses for all items; higher scores indicate higher depressive symptoms. It has been validated for use with several chronic illnesses. The PROMIS Depression Shoft Forma 6a is a common data element measurement tool that is supported by the NIH but it has not be validated with pregnant women. Therefore, we will additionally measure depressive symptoms using the Edinburgh Postnatal Depression Scale. The Edinburgh Postnatal Depression Scale is a 10-item survey questionnaire designed to detect depressive symptoms in postpartum women, with support detection of depressive symptoms in pregnancy. Scores range from 0 to 30; higher scores indicate higher depressive symptoms. We will use scores > 12 to indicate depression.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Massachusetts Amherst, Amherst, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hawkins M, Iradukunda F, Paterno M. Feasibility of a Sleep Self-Management Intervention in Pregnancy Using a Personalized Health Monitoring Device: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2019 May 29;8(5):e12455. doi: 10.2196/12455. PMID 31144670